CLINICAL TRIAL: NCT00119314
Title: Carcinoma Unknown Primary: Treatment With Gemcitabine, Docetaxel and Capecitabine (GTX) an Evaluation and Treatment Study of The Cancer Institute of New Jersey Oncology Group
Brief Title: Gemcitabine, Docetaxel, and Capecitabine in Treating Patients With Cancer of Unknown Primary Origin
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Elizabeth Poplin, MD, UMDNJ/CINJ
Organization: Rutgers, The State University of New Jersey (Other)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000433512; P30CA072720 (NIH); CINJ-000404; CINJ-4735; CINJ-NJ2203; CINJ-5073
Record Dates: First submitted 2005-07-12; First posted 2005-07-13 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2011-04

CONDITIONS: Carcinoma of Unknown Primary
Keywords: newly diagnosed carcinoma of unknown primary; recurrent carcinoma of unknown primary
MeSH Terms: conditions — Neoplasms, Unknown Primary | interventions — Capecitabine; Docetaxel; Gemcitabine; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: capecitabine
Drug: docetaxel
Drug: gemcitabine hydrochloride
Procedure: positron emission tomography

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine, docetaxel, and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving gemcitabine together with docetaxel and capecitabine works in treating patients with cancer of unknown primary origin.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the feasibility of positron emission tomography (PET) and pathology assessment in identifying the primary tumor site in patients with carcinoma of unknown primary.
* Determine the efficacy and safety of gemcitabine, docetaxel, and capecitabine in patients with carcinoma of unknown primary.

Secondary

* Determine the frequency with which PET scan and pathology assessment can define the organ of origin in these patients.

OUTLINE: This is a 2-part, multicenter study.

* Part 1: Patients undergo a comprehensive standard evaluation, including pathologic assessment and positron emission tomography scan, to attempt to identify the primary tumor site. If the primary tumor site is identified, the patient proceeds to appropriate treatment for that tumor off study. If the primary tumor site remains unknown, the patient proceeds to chemotherapy in part 2 of the study.
* Part 2: Patients receive gemcitabine IV and docetaxel IV over 30 minutes on days 4 and 11. Patients also receive oral capecitabine twice daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for 4 weeks and then every 6 months for 2 years.

PROJECTED ACCRUAL: Approximately 44 patients (10-29 for part 2) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed malignancy for which no primary origin has been identified despite routine workup, including the following:

  * History and physical examination
  * Chemistry profile and other blood work, including tumor markers with follow up on any positive findings
  * CT scan or MRI of the chest, abdomen, and pelvis
  * Mammography (for female patients)
  * Prostate examination (for male patients)
  * Stool guaiac
* Measurable disease

  * Previously irradiated lesions are not considered measurable disease unless there is documented clear tumor progression in these lesions after completion of radiotherapy
* The following tumor types or presentations are excluded:

  * Resectable disease
  * Tumors consistent with germ cell primary, as indicated by any of the following:

    * Midline tumor
    * Elevated beta human chorionic gonadotropin
    * Elevated alpha-fetoprotein
    * i12p chromosomal alteration
  * Prostate primary with elevated prostate-specific antigen
  * Females with axillary nodes as the primary disease site
  * Tumors limited to the peritoneal cavity consistent with primary peritoneal carcinoma
  * Neuroendocrine tumors
  * Squamous cell carcinoma involving cervical or inguinal lymph nodes
* No symptomatic brain metastases

  * Prior brain metastases allowed provided patient completed definitive treatment with brain irradiation with or without resection

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* More than 3 months

Hematopoietic

* Hemoglobin ≥ 9.0 g/dL
* Granulocyte count > 1,500/mm^3
* Platelet count > 100,000/mm^3

Hepatic

* Bilirubin normal
* Meets 1 of the following criteria:

  * Alkaline phosphatase (AP) normal AND AST and ALT ≤ 5 times upper limit normal (ULN)
  * AP ≤ 2.5 times ULN AND AST and ALT ≤ 1.5 times ULN
  * AP ≤ 5 times ULN AND AST and ALT normal
* Albumin ≥ 3.0 g/dL

Renal

* Creatinine ≤ 1.5 mg/dL

Gastrointestinal

* Able to take oral medication
* Intestinal absorption intact

  * No uncontrolled diarrhea and/or daily emesis

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 3 months after completion of study treatment
* No other malignancy within the past 5 years except curatively treated carcinoma in situ of the cervix or basal cell skin cancer
* No severe medical or psychiatric illness that would preclude study treatment
* No peripheral neuropathy > grade 1
* No history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for this malignancy

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* Recovered from prior radiotherapy
* Prior palliative radiotherapy to areas of bony metastases allowed provided there is measurable disease outside the radiotherapy port
* At least 4 weeks since prior radiotherapy
* No prior radiotherapy to ≥ 25% of the bone marrow

Surgery

* See Disease Characteristics

Other

* No concurrent antiviral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-07; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A. Poplin, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (6):
- United States (6):
  - Cancer Institute of New Jersey at Hamilton, Hamilton, New Jersey
  - Cancer Center at the Mountainside Hospital, Montclair, New Jersey
  - Carol G. Simon Cancer Center at Morristown Memorial Hospital, Morristown, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Hematology and Oncology Group, Somerset, New Jersey
  - Overlook Hospital, Summit, New Jersey